CLINICAL TRIAL: NCT01067495
Title: Feasibility and Effects of Cardiac Rehabilitation for Individuals After Stroke
Brief Title: Adapted Cardiac Rehabilitation After Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Dina Brooks, Toronto Rehabilitation Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSFO-SRA5977
Record Dates: First submitted 2010-02-08; First posted 2010-02-11 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; exercise; walking; risk factors
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental)
  Interventions: Behavioral: Cardiac rehabilitation

INTERVENTIONS:
Behavioral: Cardiac rehabilitation — Participants will participate in a 6-month cardiac rehabilitation exercise program. This program will include aerobic and resistance training, and education sessions on risk factor management.

SUMMARY:
Despite the similarities between heart disease and stroke in terms of disease process and elevated risk of recurrent events, exercise-based programs akin to cardiac rehabilitation are not available for people with stroke.

The purpose of this study is to examine 1) the feasibility of adapting cardiac rehabilitation for individuals with stroke, and 2) the effects of this program on aerobic capacity, walking, risk factors, community integration and quality of life.

The investigators anticipate that cardiac rehabilitation may be appropriately adapted to accommodate individuals with stroke who have a range of functional abilities, and that this program is effective in improving aerobic capacity, walking ability and stroke risk factors. The investigators also anticipate participants will demonstrate improved community integration and quality of life following this program.

DETAILED DESCRIPTION:
There are many parallels between heart disease in stroke, including their cardiovascular etiologies, presence of co-morbidities and similarities in risk factors. Cardiac rehabilitation is a well-established and successful model of care for individuals with heart disease that is focused on exercise and risk factor modification. Yet analogous secondary prevention programs for the stroke program are not readily available.

The main research question is: What is the feasibility and effect of cardiac rehabilitation in individuals following stroke?

The objectives are:

1. To determine if stroke survivors are able and willing to participate in a cardiac rehabilitation program. Specifically, to determine the feasibility of the cardiac rehabilitation program in individuals following stroke as determined by compliance to attendance and training requirements.
2. To determine if a cardiac rehabilitation program will have a meaningful benefit, among chronic stroke survivors, on:

   * walking capacity and ability: considering functional capacity [endurance / distance] and quality [neuromotor control],
   * community integration: considering quantity [activity monitors] and quality [index of reintegration to normal living] of activity
   * health-related quality of life: as determined by stroke specific index
   * risk factors for subsequent stroke: including exercise capacity, blood pressure, blood lipid profile

ELIGIBILITY:
Inclusion Criteria:

* Chedoke-McMaster Stroke Assessment (CMSA) Scale Leg Score between 3 and 7
* At least 3 months post-stroke
* Ability to understand the process and instructions for exercise training and provide informed consent
* Ability to complete 6-minute walk test

Exclusion Criteria:

* Resting blood pressure greater than 160/100 despite medication
* Other cardiovascular morbidity which would limit exercise tolerance (heart failure, abnormal blood pressure responses or ST-segment depression > 2 mm, symptomatic aortic stenosis, complex arrhythmias)
* Unstable angina
* Orthostatic blood pressure decrease of > 20 mm Hg with symptoms
* Hypertrophic cardiomyopathy
* Other musculoskeletal impairments which would limit the participant's ability to cycle or walk
* Pain or other co-morbidities (e.g. unclipped aneurysms, uncontrolled seizures etc.) which would preclude participation
* Cognitive and/or behavioural issues that would limit participation in exercise testing and training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness (aerobic capacity) and walking capacity (6 minute walk test, spatiotemporal gait parameters) | Pre-baseline (-3 months), pre-program (0 months), post-program (6 months), follow up (12 months)

SECONDARY OUTCOMES:
Plasma lipid analysis, questionnaires pertaining to quality of life and community integration | Pre-baseline (-3 months), pre-program (0 months), post-program (6 months), follow up (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: William E McIlroy, PhD, Principal Investigator — University of Waterloo; Paul Oh, MD, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute Cardiac Rehabilitation and Secondary Prevention Program - Rumsey Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Tang A, Marzolini S, Oh P, McIlroy WE, Brooks D. Feasibility and effects of adapted cardiac rehabilitation after stroke: a prospective trial. BMC Neurol. 2010 Jun 9;10:40. doi: 10.1186/1471-2377-10-40. PMID 20529376